CLINICAL TRIAL: NCT02642978
Title: The Safety and Effect of Robot-assisted Procedure Versus Open Simultaneous Resection of Colorectal Cancer： Randomized Control Trial Study
Brief Title: Robot-assisted Procedure Versus Open Simultaneous Resection of Colorectal Cancer With Liver Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xu jianmin (Other)
Responsible Party: Sponsor-Investigator, Xu jianmin, Fudan University, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSRCLM
Record Dates: First submitted 2015-09-08; First posted 2015-12-30 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Liver Metastasis
Keywords: minimally invasive surgery; colorectal liver metastasis; robotic surgery; Patients with resectable colorectal liver metastasis

STUDY DESIGN:
Intervention Model Description: micro-invasive surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RSRCLM (Experimental): robot-assisted, simultaneous radical resection of both colorectal cancer and liver metastasis (RSRCLM).Three different liver resection procedures were chose to personalized patients. Generally, when the size of liver metastasis was ≤ 3 cm, a wedge resection was chose without Hilar vessels blocking. The segmentectomy was performed using the Glissonian approach when tumor size was among 3-5 cm, and Hilar vessels was blocked, if necessary. For resection of Couinaud's segments II and III, left lateral sectionectomy (LLS) was performed commonly. Intraoperative ultrasound can help us find intrahepatic pedicles and follow the proper resection line. When liver tumor size was more than 5 cm or more than 3 tumors with the size over 3cm, hemicolectomy was applied usually.
  Interventions: Procedure: RSRCLM
- Open (Active Comparator): Traditional open simultaneous radical resection of both colorectal cancer and liver metastasis. The DFS and safety event were evaluated.
  Interventions: Procedure: Open

INTERVENTIONS:
Procedure: RSRCLM — The Da Vinci Surgical System may help to overcome some of the difficulties of laparoscopy for complicated abdominal surgery. The aim of this study was to present an innovative technique that is robot-assisted, simultaneous radical resection of both colorectal cancer and liver metastasis (RSRCLM).
  Arms: RSRCLM
Procedure: Open — Traditional open simultaneous radical resection of both colorectal cancer and liver metastasis
  Arms: Open

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of robot-assisted simultaneous resection in selected patients with sigmoid colon cancer or rectal cancer liver metastases, and compared with the traditional open procedure.

DETAILED DESCRIPTION:
The Da Vinci Surgical System may help to overcome some of the difficulties of laparoscopy for complicated abdominal surgery. The aim of this study was to present an innovative technique that is robot-assisted, simultaneous radical resection of both colorectal cancer and liver metastasis (RSRCLM).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years;
2. Primary tumor has undergone histologically confirmed colon adenocarcinoma; Colon cancer was defined by the presence of the inferior pole of the tumor above the peritoneal reflection (at least 15 cm from the anal margin).
3. Together with clinical or radiological evidence of Stage II (T3-4, N0, M0) or Stage III (T1-4, N1-2, M0) disease (according to the 2010 revision of the International Union Against Cancer primary tumor, regional nodes, metastasis (TNM) staging system);Liver metastasis was diagnosis by multidisciplinary (MDT) team base on liver Magnetic Resonance Imaging (MRI) and Positron Emission Computed Tomography (PET-CT).
4. Performance status (ECOG) 0~1
5. Adequate hematological function: Neutrophils≥1.5 x109/l and platelet count≥100 x109/l; hemoglobin (Hb) ≥9g/dl (within 1 week prior to randomization)
6. Adequate hepatic and renal function: Serum bilirubin≤1.5 x upper limit of normal (ULN), alkaline phosphatase ≤5x ULN, and serum transaminase (either primary tumor, regional nodes, metastasis (AST) or ALT) ≤ 5 x ULN(within 1 week prior to randomization);
7. Written informed consent for participation in the trial.
8. The liver resectability was evaluated by liver surgery of MDT team, indication including: tumor number ≤ 3; the Maximum diameter of one tumor ≤ 10 cm.

Exclusion Criteria:

1. Body mass index (BMI) more than 30 kg/m2.
2. Serious pre-operative comorbidity, including cardiovascular disease (coronary arteriosclerosis, arrhythmia, heart failure), pulmonary dysfunction (lung emphysema, obstructive lung disease), liver insufficiency (Child-Pugh B or C), renal insufficiency (serum creatinine >2.0 mg/dl), and arterial circulation disturbance (occlusion of arterial vessels of limb in patient's history.
3. History of accepting abdominal surgery.
4. Liver tumor located at I or invasive the middle hepatic vein.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Surgical Complication | 30 days after surgury
  According to Clavein-Dindo complication system to calculate the complication events during 30 day after surgery

SECONDARY OUTCOMES:
Operative mortality | 30 days post operatively
  death occurred 30 days after operation
Disease-free survival(DFS) | 3 years disease-free survival
  DFS was defined as from the date of randomization to the date of tumor
overall survival (OS) | OS rate at 3 and 5 years after operation
  overall survival was defined as from the date of randomization to the date of Death ;
locoregional recurrence rate | 3 and 5 years
  local recurrence rate at 3 and 5 years after operation

OTHER OUTCOMES:
self reported bladder function | at postoperative 3, 6 and 1 2 months
  This section is assessed using a self-rating scale "International prostate symptom score" (IPSS)
self reported sexual function for male patients | at postoperative 3, 6 and 1 2 month
  This section is assessed using a self-rating scale "International Index of Erectile Function" (IIEF-5).
self reported sexual function for female patients | at postoperative 3, 6 and 1 2 months
  This section is assessed using a self-rating scale "Female Sexual Function Index" (FSFI).
liver function | at Day 1，3，5 after surgery
  Serum aminotransferase will be tested in the laboratory

CONTACTS AND LOCATIONS:
Overall Officials: wenju chang, MD, Principal Investigator — Fudan University
Locations (1):
- Department of General Surgery, Zhongshan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang W, Ye Q, Xu D, Liu Y, Zhou S, Ren L, He G, Zhou G, Liang F, Fan J, Wei Y, Wang X, Xu J. Robotic versus open surgery for simultaneous resection of rectal cancer and liver metastases: a randomized controlled trial. Int J Surg. 2023 Nov 1;109(11):3346-3353. doi: 10.1097/JS9.0000000000000581. PMID 37800563